CLINICAL TRIAL: NCT01547702
Title: Randomized-controlled Trial of a Classroom-based Distance Intervention for Teachers of Elementary School-aged Children With ADHD
Brief Title: Classroom-based Distance Intervention for Teachers of Children With Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dalhousie University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSHRF-44576
Record Dates: First submitted 2012-02-27; First posted 2012-03-08 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: ADHD; attention; inattention; hyperactivity; classroom intervention; teacher education; web-based intervention
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): This group will have access to the Teacher Help for ADHD intervention program during the randomized controlled trial.
  Interventions: Behavioral: Teacher Help for ADHD
- Waitlist Control (No Intervention): This group will not receive the intervention until all data collection is complete for their study cohort.

INTERVENTIONS:
Behavioral: Teacher Help for ADHD — Teachers will review powerpoints other materials online and will have access to a study coach to assist with their understanding and practical application of the materials. Session descriptions follow:
  * Session 1: Provide information about ADHD characteristics, impact, diagnosis, etiology
  * Session 2: Help establish teacher's role; goal setting; introduce behaviour planning
  * Session 3: Help develop and implement behaviour program specific to the needs of students with Session 2 goals
  * Session 4: Help develop strategies re: classroom structure, work assignments, teacher-student relationship
  * Session 5: Help to use instructional interventions for ADHD
  * Session 6: Help to teach these students self-monitoring and self-evaluation skills; help teachers to evaluate progress, phase out behaviour program, and plan for relapses in unwanted behaviours
  Arms: Treatment

SUMMARY:
The purpose of this study is to evaluate, by way of randomized controlled trial, the effectiveness of a web-based, time-flexible, and teacher-directed "Teacher Help for ADHD" program in reducing the impact of ADHD symptoms in elementary students.

DETAILED DESCRIPTION:
*Please note that the information below is taken verbatim from our project's research summary.*

Treatment of Attention-Deficit/Hyperactivity Disorder (ADHD) is one of the most well-researched areas in childhood psychopathology. ADHD is a highly prevalent (5% of school-aged children) and chronic disorder (ADHD will persist into adulthood for ~70% of children diagnosed with this disorder). ADHD has a substantial impact on daily life including difficulties with behavioural, academic, social and emotional functioning (DuPaul & Weyandt, 2006).

Although medication is the most commonly used treatment, there are a number of important limitations including poor long-term effects, lack of effectiveness in improving academic skills, and lack of acceptability by parents and children (DuPaul, 2007). Therefore, a number of psychosocial interventions have been developed and empirically validated (parent training, social skills training, school-based interventions). School-based interventions have been shown to be effective; however, these are significantly underutilized and when implemented in an uncontrolled way, are often ineffective. This intervention program is comprised of evidence-based treatment strategies that are presented in a manner that will provide teachers with knowledge of the disorder and intervention strategies. The novel delivery of this program, through distance treatment modalities (e-mail and internet) will allow us to overcome many of the known barriers to treatment so that teachers will receive the necessary information in a timely and efficient manner. The specific research questions that will be addressed are:

1. Does the overall impairment of children with ADHD in the treatment group improve compared to those who are in the waitlist group?
2. Is the school-based intervention effective in reducing ADHD symptoms, improving behavioral functioning, and enhancing academic performance in the active treatment group compared to the waitlist group?
3. Do teachers in the treatment group develop more knowledge about ADHD and more positive and realistic attitudes about this disorder over the course of the intervention?
4. Is the intervention viewed as accessible to teachers and is there evidence of fidelity to the program?

The investigators expect that the program will reduce overall impairment, improve ADHD symptoms, behavioural, and academic functioning in the children and will enhance knowledge and reduce misconceptions of ADHD in teachers. If successful, this program will be disseminated to school boards in Nova Scotia and across Canada, and as such would have the potential to have a significant positive effect on the health and well-being of many children, teachers and parents.

ELIGIBILITY:
Inclusion Criteria:

* Student is in grades 1 to 6 in the public school English stream
* Student has been formally diagnosed with Attention Deficit Hyperactivity Disorder having a diagnosis of ADHD
* Student is either on a stable dose of medication or no medication with no plan to start/change medication in the next 5 months

Exclusion Criteria:

* Student has a significant other mental health issue (e.g., depression, anxiety, suicidal ideation, psychotic features, and severe conduct problems)
* Student is on an Individualized Program Plan (IPP) due to significant physical, behavioural, communication, or learning difficulties.
* Teacher participated in the Teacher Help for ADHD pilot study (conducted by Brittany Barnett, Master of Health Informatics Student under the supervision of Dr. Elik and Dr. Corkum, Dalhousie University)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2012-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The Impairment Rating Scale (IRS, Fabiano & Pelham, 2002) | Change from Baseline in ADHD symptom impairment at 6 weeks (length of intervention) and 12 weeks (follow-up)
  The IRS will be the primary outcome measure in our study because it assesses the areas of functioning that are impacted most by the symptoms of ADHD. It consists of six questions on the teacher version and seven questions on the parent version, which measure the child's academic, behavioural, relational functioning and self-esteem.

SECONDARY OUTCOMES:
Knowledge of Attention Deficit Disorder Scale (KADDS; Sciutto, Terjesen, & Bender, 2000) | Change from Baseline in ADHD knowledge at 6 weeks (length of intervention) and 12 weeks (follow-up)
  The KADDS is 36-item True/False questionnaire used to evaluate parents' and teachers' ADHD knowledge. Parents will complete this only at baseline, while teachers will be asked to complete it during baseline, end of trial, and follow up data collection periods.
Beliefs about Attention Deficit Hyperactivity Disorder (Kos, 2008) | Change from Baseline in ADHD beliefs at 6 weeks (length of intervention) and 12 weeks (follow-up)
  This is a 31-item scale used to evaluated attitudes and beliefs about ADHD. Parents/teachers are asked to indicate on a 5-point scale (ranging from Strongly Agree to Strongly Disagree) how much they agree with various statements about ADHD. Parents will complete this only at baseline, while teachers will be asked to complete it during baseline, end of trial, and follow up data collection periods.
Instructional and Behavior Management Approaches Survey (IBMA; Martinussen, Tannock, & Chaban, 2011) | Change from Baseline in behaviour management approaches at 6 weeks (length of intervention) and 12 weeks (follow-up)
  The IBMA is a 40-item scale used to evaluate teacher's classroom management practices. Teachers are asked to indicate on a 5-point scale (ranging from Rarely to Most of the time) how often they use the listed behavioural strategies.
Intention and Subjective Norm questionnaires (Based on Prochaska & DiClemente's Stages of Change Model, 1984) | Change from Baseline in intentions and subjective norms at 6 weeks (length of intervention) and 12 weeks (follow-up)
  These brief questionnaires contain 5 items in total and are used to evaluate teachers' intention to change and external sources of motivation as related to learning more about ADHD.
Swanson, Kotkin, Agler, M-Flynn, and Pelham Scale (SKAMP; see Murray, Bussing, Fernandez, Hou, Garvan, Swanson, & Eyberg, 2009) | Functional impairment of ADHD symptoms will be measured in the Treatment group at 2 weeks, 3 weeks, 4 weeks, 5 weeks, 6 weeks, and 7 weeks
  The SKAMP is a 10-item questionnaire that measures the functional impairment of ADHD symptoms in the school setting. Statements target children's classroom attention and deportment, and teachers are asked to respond on a 4-point Likert-type scale, response items ranging from "Not at All" to "Very much."
Homework Problem Checklist (HPC; Anesko, Schoiock, Ramirez, & Levine, 1987) | Change from Baseline in homework problems at 6 weeks (length of program) and 12 weeks (follow-up)
  The HPC is a parent report instrument consisting of 20 items. It has been used in a number of studies as a screening tool and outcome measure to assess homework problems.
Parent and Teacher Satisfaction Ratings (adapted from Ervin, DuPaul, Kern, & Friman, 1998) | Treatment group will complete satisfaction questionnaires at 6 weeks
  Two versions of this questionnaire are used to assess parent and teacher satisfaction with interventions for children with ADHD. The parent version consists of 10 items and the teacher version consists of 15 items, rated on an 6-point Likert scale ranging from 1 (strongly disagree) to 6 (strongly agree). Items focused on intervention effectiveness (e.g., ''problem behavior improved during the intervention''), feasibility (e.g., ''the intervention was easy to implement''), and social validity (e.g., ''the student seemed to appreciate the intervention'').
Conners 3rd Edition Parent and Teacher Rating Scales (Full-length) (Conners 3-P, Conners 3-T; Conners, 2008) | Change from Baseline in problem behaviours at 6 weeks (length of program) and 12 weeks (follow-up)
  The Conners 3-P and Conners 3-T are a 110-item and 115-item behavior rating scale designed to evaluate problem behaviors in the home and school settings in children aged 6 to 18 years.. These measures are the most widely used measures of ADHD symptoms in treatment trials. These measures will be accessed through a secure web link.
Home & School Situations Questionnaire (HSQ/SSQ; Barkley & Murphy, 2005) | Change from Baseline in behaviours at 6 weeks (length of program) and 12 weeks (follow-up)
  The HSQ and SSQ evaluate the pervasiveness of children's behaviour problems in the home and school setting. Parents/Teachers are asked to rate their child's/student's behaviour problems across 16 different home/school situations using a 9-point Likert scale (1=mild to 9=severe).
Academic Performance Rating Scale (APRS; DuPaul, Rapport, & Perriello, 1991) | Change from Baseline in academic performance at 6 weeks (length of program) and 12 weeks (follow-up)
  The APRS is a 19-item questionnaire that measures academic accuracy and productivity in the classroom. Factor analysis resulted in four scales (Total score, Academic Success, Impulse Control, and Academic Productivity). All scales will be used in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Penny V Corkum, PhD, Principal Investigator — Dalhousie University; Nezihe Elik, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Dalhousie University, Halifax, Nova Scotia, Canada